CLINICAL TRIAL: NCT05796440
Title: An Extension Study to Monitor Long-Term Safety of LUM-201 Treatment in Children With Idiopathic Growth Hormone Deficiency
Brief Title: A Long-Term Safety Trial of LUM-201 in Children With Idiopathic Growth Hormone Deficiency Who Have Previously Completed a LUM-201 Clinical Trial (OraGrowtH211)
Acronym: OraGrowtH211
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Lumos Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-201-02
Record Dates: First submitted 2023-03-19; First posted 2023-04-03 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Growth Hormone Deficiency
Keywords: LUM-201; PGHD; GHD; Growth hormone secretagogue; Oral; Height
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LUM-201 (1.6 mg/kg/day) (Experimental)
  Interventions: Drug: LUM-201

INTERVENTIONS:
Drug: LUM-201 — Administered orally once daily

SUMMARY:
This is a multi-national trial. The trial aims to study the long-term safety of LUM-201 in subjects with Idiopathic Pediatric Growth Hormone Deficiency (iPGHD). This study will also assess pharmacodynamics and efficacy response to therapy with LUM-201.

DETAILED DESCRIPTION:
An Extension Study to Monitor Long-Term Safety of LUM-201 Treatment in Children with Idiopathic Growth Hormone Deficiency. This study will last for up to 36 months to allow collection of additional long-term safety and efficacy data related to LUM-201 treatment in the pediatric patient population. Subjects will enter into this trial after successful participation in a prior LUM-201 study. This study will consist of visits every 6 months through three years.

There are a total of 7 in-person visits with a follow-up phone call between visits. At the clinic visits, subjects will have a physical exam and blood collection as well as efficacy assessments.

ELIGIBILITY:
Inclusion Criteria:

* Parent/caregiver must sign the informed consent, and the subject must sign the assent, as applicable.
* Must have successfully participated in a pediatric LUM-201 GHD study through at least the 12-month visit, and be eligible for continuation of treatment, pending all other enrollment criteria are met.

Exclusion Criteria:

* Medical or genetic condition that, in the opinion of the PI and/or MMs, adds unwarranted risk to the use of LUM-201
* Has planned or is receiving current long-term treatment with medications known to act as substrates, inducers, or inhibitors of the cytochrome system CYP3A4 that metabolizes LUM-201. Subjects receiving shorter-term (two weeks or less) treatment with these medications should be evaluated on case-by-case basis by the PI in consultation with the MMs.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Day 1 to Month 36
  Number of events

SECONDARY OUTCOMES:
Growth Hormone Concentrations in subjects | Day 1 to Month 36
  Serum GH concentration
Insulin-like growth factor 1 concentration | Day 1 to Month 36
  Serum concentrations of insulin-like growth factor 1
Height standard deviation score (SDS) | Day 1 to Month 36
  Change in HT-SDS
Change in Weight SDS | Day 1 to Month 36
  Change in Weight
Annualized Height Velocity (AHV) achieved by daily dosing 1.6mg/kg of LUM-201 | Day 1 to Month 36
  (AHV) measured as standing height with stadiometer
Change in Bone Age (BA) | Day 1 to Month 36
  Change in Bone Age (BA) compared to Chronological Age

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - University of Iowa, Iowa City, Iowa
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of South Carolina, Charleston, South Carolina
  - Texas Tech University Health Sciences Center, Amarillo, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Canberra Hospital, Garran, Australian Capital Territory, Australia